CLINICAL TRIAL: NCT02673034
Title: Circadian Variation in Serum-progesterone Levels Following Controlled Ovarian Hyperstimulation.
Status: Completed | Type: Observational
Sponsor: Regionshospitalet Viborg, Skive (Other)
Responsible Party: Principal Investigator, Peter Humaidan, Professor, DMSc, Regionshospitalet Viborg, Skive
Other Study IDs: CirProg
Record Dates: First submitted 2016-02-01; First posted 2016-02-03 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of the study is to investigate the circadian variation in serum-progesterone in women undergoing controlled ovarian stimulation.

ELIGIBILITY:
Inclusion Criteria:

Women undergoing standard IVF/ICSI treatment.

Exclusion Criteria:

Previous participation in the study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women undergoing IVF-treatment using either GnRHa long protocol or GnRH antagoinst co-treatment.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
serum progesterone levels | 12 hours

SECONDARY OUTCOMES:
serum LH levels | 12 hours
serum estradiol levels | 12 hours
17-OH progesterone | 12-hours

CONTACTS AND LOCATIONS:
Locations (1):
- The Fertility Clinic Skive, Skive, Resenvej 25, Denmark

IPD SHARING:
Plan to Share IPD: No